CLINICAL TRIAL: NCT06148675
Title: MINT Registry : Macrowire for IntracraNial Thrombectomy
Brief Title: Macrowire for IntracraNial Thrombectomy
Acronym: MINT
Status: Completed | Type: Observational
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Kaustubh Limaye, Assistant Clinical Professor Of Neurology, Neurological Surgery and Radiology, Indiana University
Other Study IDs: 19347
Record Dates: First submitted 2023-11-20; First posted 2023-11-28 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Stroke, Acute Ischemic
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants with emergent large vessel occlusion undegoing intracranial mechanical thromebctomy: Participants with emergent large vessel occlusion undergoing intracranial mechanical thrombectomy where the reperfusion catheter was delivered over a macrowire to perform thrombectomy.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — No intervention,data collection

SUMMARY:
The aim of this study is to develop a multicenter database of patient data and outcomes for patients undergoing intracranial thrombectomy for acute ischemic stroke secondary to emergent large vessel occlusion with delivery of reperfusion catheter over a novel macrowire (Aristotle Colossus) to perform intracranial mechanical thrombectomy.

ELIGIBILITY:
Inclusion Criteria:

Age >18-85 years Time of onset < 24 hours Acute stroke patient with NIHSS >6 CT-ASPECTS ≥ 6 Proven intracranial occlusion - (ICA-T, M1) Modified Rankin score: 0-2

Exclusion Criteria:

Age <18 years or >85 years Unknown time of onset NIHSS < 5 CT ASPECTS <5 Pre-stroke morbidity, modified Rankin score > 2 Tandem occlusion

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects aged 18-85 years will be identified once they undergo mechanical thrombectomy for large vessel occlusion where delivery of reperfusion catheter over macrowire alone was performed.
Sampling Method: Non-Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2023-05-25 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
Ability to deliver reperfusion catheter to the intracranial occlusion with macrowire alone (Yes/No) | Intraprocedure

SECONDARY OUTCOMES:
Time from vascular access to first intracranial pass (minutes) | Procedure duration
Time from vascular access to recanalization (minutes) | Procedure duration
Vessel dissection (Yes/No) | Intraprocedure

CONTACTS AND LOCATIONS:
Overall Officials: Kaustubh Limaye, MD, Principal Investigator — Indiana University
Locations (1):
- Indiana University Methodist Hospital, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No
All data will be de-identified

REFERENCES:
- [Background] Berkhemer OA, Fransen PS, Beumer D, van den Berg LA, Lingsma HF, Yoo AJ, Schonewille WJ, Vos JA, Nederkoorn PJ, Wermer MJ, van Walderveen MA, Staals J, Hofmeijer J, van Oostayen JA, Lycklama a Nijeholt GJ, Boiten J, Brouwer PA, Emmer BJ, de Bruijn SF, van Dijk LC, Kappelle LJ, Lo RH, van Dijk EJ, de Vries J, de Kort PL, van Rooij WJ, van den Berg JS, van Hasselt BA, Aerden LA, Dallinga RJ, Visser MC, Bot JC, Vroomen PC, Eshghi O, Schreuder TH, Heijboer RJ, Keizer K, Tielbeek AV, den Hertog HM, Gerrits DG, van den Berg-Vos RM, Karas GB, Steyerberg EW, Flach HZ, Marquering HA, Sprengers ME, Jenniskens SF, Beenen LF, van den Berg R, Koudstaal PJ, van Zwam WH, Roos YB, van der Lugt A, van Oostenbrugge RJ, Majoie CB, Dippel DW; MR CLEAN Investigators. A randomized trial of intraarterial treatment for acute ischemic stroke. N Engl J Med. 2015 Jan 1;372(1):11-20. doi: 10.1056/NEJMoa1411587. Epub 2014 Dec 17. PMID 25517348
- [Background] Goyal M, Demchuk AM, Menon BK, Eesa M, Rempel JL, Thornton J, Roy D, Jovin TG, Willinsky RA, Sapkota BL, Dowlatshahi D, Frei DF, Kamal NR, Montanera WJ, Poppe AY, Ryckborst KJ, Silver FL, Shuaib A, Tampieri D, Williams D, Bang OY, Baxter BW, Burns PA, Choe H, Heo JH, Holmstedt CA, Jankowitz B, Kelly M, Linares G, Mandzia JL, Shankar J, Sohn SI, Swartz RH, Barber PA, Coutts SB, Smith EE, Morrish WF, Weill A, Subramaniam S, Mitha AP, Wong JH, Lowerison MW, Sajobi TT, Hill MD; ESCAPE Trial Investigators. Randomized assessment of rapid endovascular treatment of ischemic stroke. N Engl J Med. 2015 Mar 12;372(11):1019-30. doi: 10.1056/NEJMoa1414905. Epub 2015 Feb 11. PMID 25671798
- [Background] Albers GW, Lansberg MG, Kemp S, Tsai JP, Lavori P, Christensen S, Mlynash M, Kim S, Hamilton S, Yeatts SD, Palesch Y, Bammer R, Broderick J, Marks MP. A multicenter randomized controlled trial of endovascular therapy following imaging evaluation for ischemic stroke (DEFUSE 3). Int J Stroke. 2017 Oct;12(8):896-905. doi: 10.1177/1747493017701147. Epub 2017 Mar 24. PMID 28946832
- [Background] Turk AS, Frei D, Fiorella D, Mocco J, Baxter B, Siddiqui A, Spiotta A, Mokin M, Dewan M, Quarfordt S, Battenhouse H, Turner R, Chaudry I. ADAPT FAST study: a direct aspiration first pass technique for acute stroke thrombectomy. J Neurointerv Surg. 2018 Jul;10(Suppl 1):i4-i7. doi: 10.1136/neurintsurg-2014-011125.rep. PMID 30037944
- [Background] Hesse AC, Behme D, Kemmling A, Zapf A, Grosse Hokamp N, Frischmuth I, Maier I, Liman J, Tsogkas I, Buhk JH, Tran J, Fiehler J, Mpotsaris A, Schramm P, Berlis A, Knauth M, Psychogios MN. Comparing different thrombectomy techniques in five large-volume centers: a 'real world' observational study. J Neurointerv Surg. 2018 Jun;10(6):525-529. doi: 10.1136/neurintsurg-2017-013394. Epub 2017 Sep 28. PMID 28963362
- [Background] Heit JJ, Wong JH, Mofaff AM, Telischak NA, Dodd RL, Marks MP, Do HM. Sofia intermediate catheter and the SNAKE technique: safety and efficacy of the Sofia catheter without guidewire or microcatheter construct. J Neurointerv Surg. 2018 Apr;10(4):401-406. doi: 10.1136/neurintsurg-2017-013256. Epub 2017 Aug 2. PMID 28768818